CLINICAL TRIAL: NCT02535819
Title: Endothelial Cell Loss After Phacoemulsification Intra and Supracapsular
Acronym: PERCEPOLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-01-CHRMT; 2015-A00789-40 (Other: ANSM)
Record Dates: First submitted 2015-06-30; First posted 2015-08-31 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2017-09

CONDITIONS: Cataracts
Keywords: Cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subluxation (Experimental): Nucleus is hydrodissected until it lilts above the capsular bag, rotated to face the incision then tumbled and emulsification continues from the opposite equator outside in until complete
  Interventions: Procedure: Subluxation
- Divide and Conquer (Other): Cataract nucleus is fragmented into 4 pieces then aspirated by ultrasonic vibration
  Interventions: Procedure: Divide and Conquer

INTERVENTIONS:
Procedure: Subluxation — One pole of The nucleus is hydrodissected until it lilts above the capsular bag. The tilted nucleus is rotated to face the incision and remaining half nucleus is then tumbled and emulsification continues from the opposite equator outside in until complete
  Arms: Subluxation
Procedure: Divide and Conquer — Cataract nucleus is fragmented into 4 pieces then aspirated by ultrasonic vibration
  Arms: Divide and Conquer

SUMMARY:
Cataract is the clouding of the lens of the eye, which initially prevents clear vision and eventually progresses to blindness if left untreated. Cataract remains the leading cause of blindness and an important cause of visual impairment across the globe. Cataract surgery by ultrasonic phacoemulsification is the most common surgery practiced in France (600 000/year)

Two sub-categories of phacoemulsification coexist :

Endocapsulars techniques represented by Divide-and-Conquer and Phaco-Chop ; and Supracapsular techniques mainly represented by Subluxation (similar to Tilt-and-Tumble) The corneal endothelium plays an important role in maintaining the dehydrated state and the transparency of the cornea. Some degree of endothelial cell loss invariably occurs in all types of cataract surgery but the amount of endothelial cell loss may varies with the type of surgical technique The aim of the study is to evaluate the density of the central corneal endothelial cells before and after cataract surgery comparing two phacoemulsification techniques (Divide-and-Conquer vs Subluxation)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Patients undergoing cataract surgery
* Visual acuity Monoyer scale <6/10e (< +0.2 logMar)
* Nuclear, cortical and posterior subcapsular cataract with normal density to severe in the LOCSIII classification

Exclusion Criteria:

* insulin-dependent diabetes and /or diabetic retinopathy
* corneal disease: keratitis, dystrophy, corneal degeneration
* Any disease of intraocular pressure
* Any disease of the anterior segment
* Low preoperative endothelial cell density < 1500 c/mm²
* Combined surgery (cataract + corneal transplant, cataract + glaucoma surgery, cataract +vitrectomy ...)
* Risk factors for surgical per-operative complication
* Pregnancy, lactation
* Ward of court
* Patient not covered by the Social Security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Main Outcome Measures: postoperative Endothelial cell loss of the central corneal | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERONE, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- Chr Metz Thionville, Metz, France

REFERENCES:
- [Derived] Leterrier J, Mastrangelo L, Goetz C, Zevering Y, Perone JM. Preoperative and perioperative factors that predict endothelial cell loss 1 year after uncomplicated Descemet membrane endothelial keratoplasty. PLoS One. 2025 Dec 19;20(12):e0339346. doi: 10.1371/journal.pone.0339346. eCollection 2025. PMID 41417772
- [Derived] Perone JM, Ghetemme C, Zevering Y, Zaidi M, Ouamara N, Goetz C, Lhuillier L. Corneal Endothelial Cell Loss After Endocapsular and Supracapsular Phacoemulsification: The PERCEPOLIS Randomized Clinical Trial. Cornea. 2022 Jun 1;41(6):714-721. doi: 10.1097/ICO.0000000000002822. Epub 2021 Nov 2. PMID 34732666